CLINICAL TRIAL: NCT06053957
Title: The Effect of Early Mobilization on Postoperative Recovery in Abdominal Surgery: A Randomized Controlled Study
Brief Title: The Effect of Early Mobilization on Postoperative Recovery in Abdominal Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cumhuriyet University (Other)
Responsible Party: Principal Investigator, Kubra Erturhan Turk, Assistant Prof, Cumhuriyet University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CumhuriyetTURK01
Record Dates: First submitted 2023-09-17; First posted 2023-09-26 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-05

CONDITIONS: Nursing Caries; Early Ambulation
Keywords: Early ambulation; abdominal surgery; nursing; postoperative recovery
MeSH Terms: interventions — Early Ambulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mobilization (Experimental): Patients undergoing early mobilization program
  Interventions: Procedure: early mobilization
- mobilization free (No Intervention): Patients not subjected to early mobilization program

INTERVENTIONS:
Procedure: early mobilization — early mobilization program
  Arms: Mobilization

SUMMARY:
Objectives: This study will be conducted to determine the effect of early mobilization on postoperative recovery in abdominal surgery patients..

Methods: This research is a randomized controlled experimental study. In the Gastrointestinal Surgery Department, a total of 130 patients will be included, consisting of 65 experimental group and 65 control group, who are scheduled for abdominal surgery in the study. In the study, data will be collected using a survey form, Numerical Rating Scale, gradual mobilization chart in the first 24 hours after surgery, and Postoperative Recovery Index (PoRI-TR). On the day before the surgery, the experimental group will receive early mobilization training. On the day of the surgery, vital signs, oxygen saturation, and pain intensity will be assessed before the first mobilization. Pain control will be ensured before mobilization. Each mobilization will be carried out in accordance with the gradual mobilization schedule within the first 24 hours after surgery. Following the Enhanced Recovery After Surgery (ERAS) protocol recommendation, mobilization will be provided outside of bed for a total of 2 hours, with durations increasing by the hour on the day of surgery under the supervision of the researcher: 5, 15, 25, 35, and 40 minutes. Mobilizations for patients showing signs of orthostatic hypotension will be postponed by 30 minutes. On the days following the surgery, patients will be informed to spend 6 hours outside of bed. The control group will receive routine care procedures. The second part of the questionnaire will be administered on the day of the surgery for both the experimental and control groups, and the PoRI-TR will be applied at the 25th hour after surgery. Data will be collected through face-to-face interviews within 20-25 minutes. The data obtained from the research will be evaluated using the SPSS 22.00 program. The normality of the data will be determined by Skewness-Kurtosis tests. Based on this result, either parametric or non-parametric tests will be applied.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are conscious,
* Without cognitive or mental problems,
* Undergoing elective abdominal surgery,
* Aged 18 and above,
* Without physical limitations preventing early mobilization,
* Without active bleeding,
* Without cardiovascular or respiratory diseases,
* Classified as American Society of Anesthesiologists (ASA) class I or II,
* Literate patients
* Volunteering

Exclusion criteria:

* Patients undergoing oncologic surgery who spend the first 24 hours in the intensive care unit due to post-operative care,
* Emergency surgery patients due to the absence of pre-operative preparation phase,
* Patients who are healthcare workers due to their knowledge about early mobilization

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2023-09-16 (Actual); Primary Completion 2024-01-29 (Actual); Study Completion 2024-02-29 (Actual)

PRIMARY OUTCOMES:
The time to start the first mobilization | The time of the first mobilization within the first 24 hours after the surgery will be recorded.
Postoperative recovery index results | The postoperative recovery index will be applied at the 24th hour.
Total mobilization time in the first 24 hours | Total mobilization time will be applied at the 24th hour.

CONTACTS AND LOCATIONS:
Locations (1):
- Kubra Erturhan Turk, Sivas, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No